CLINICAL TRIAL: NCT00696163
Title: A Multicentre, Open Label, Nonrandomised, Non- Interventional, A Multicentre, Open Label, Nonrandomised, Non- Interventional, Observational Study to Evaluate the Quality of Life and Clinical Outcomes in Subjects Using Biphasic Insulin Aspart 30 (NovoMix® 30) for the Treatment of Diabetes Mellitus
Brief Title: Observational Study to Assess the Quality of Life and Clinical Outcomes in Subjects Using NovoMix® 30 for the Treatment of Diabetes
Acronym: IMPROVE Life
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: BIASP-3555
Record Dates: First submitted 2008-06-10; First posted 2008-06-12 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: biphasic insulin aspart 30

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — Being an observational study, dose of NovoMix 30 will be according to treating physician's discretion
  Other Names: NovoMix® 30; BIAsp30

SUMMARY:
This study is conducted in Asia. The aim of this observational study is to evaluate the quality of life and clinical outcomes in subjects using NovoMix® 30 (biphasic insulin aspart 30) for the treatment of diabetes mellitus under normal clinical practice conditions in India.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes, including newly-diagnosed who have never received insulin or an insulin analogue before, at the discretion of the physician.

Exclusion Criteria:

* Currently treated with NovoMix® 30
* Subjects who are unlikely to comply with protocol requirements
* Previously enrolled in this study
* Hypersensitivity to biphasic insulin aspart or to any of the excipients
* Women who are pregnant, breast feeding or have the intention of becoming pregnant within next 12 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Type 2 diabetes
Sampling Method: Probability Sample
Enrollment: 24975 (Actual)
Dates: Start 2008-04; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Change in Quality of Life from baseline (using QoLD questionnaire) | From baseline to 26 weeks of treatment

SECONDARY OUTCOMES:
Safety | After 26 weeks
Efficacy | After 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Bangalore, India

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com